CLINICAL TRIAL: NCT00739206
Title: A Multicenter, Open Label, Efficacy and Safety Study of Parenteral SAR97276A in the Treatment of Symptomatic Uncomplicated and Severe Malaria in Adults and Children
Brief Title: Study of SAR97276A in the Treatment of Uncomplicated and Severe Malaria in Adults and Children.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In accordance with protocol's predefined criteria and Data Monitoring Committee recommendation due to insufficient level of efficacy
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT10004
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Malaria
Keywords: uncomplicated; severe; treatment; Plasmodium Falciparum
MeSH Terms: conditions — Malaria; Lymphoma, Follicular; Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): Adult patients with uncomplicated malaria
  Interventions: Drug: SAR97276A
- Cohort 2 (Experimental): Pediatric patients with uncomplicated malaria
  Interventions: Drug: SAR97276A
- Cohort 3 (Experimental): Pediatric patients with severe malaria
  Interventions: Drug: SAR97276A

INTERVENTIONS:
Drug: SAR97276A — Dose based on body weight

SUMMARY:
The objective of the study is to assess the efficacy and safety of SAR97276A in severe malaria in pediatric patients. Before treating pediatric patients with severe malaria, the efficacy and safety of SAR97276A will be first tested in adult patients, then in pediatric patients, with uncomplicated malaria.

The safety and the concentration of SAR97276A in blood and plasma will be assessed in adult and pediatric patients.

DETAILED DESCRIPTION:
The treatment will be administered by intramuscular or intravenous route depending on the cohort. The treatment will be administered as single dose or 3-day repeated dose. The patients will be hospitalized for 3 days and followed up to 28 days following study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with uncomplicated malaria will be enrolled in cohort 1
* Pediatric patients with uncomplicated malaria will be enrolled in cohort 2
* Pediatric patients with severe malaria will be enrolled in cohort 3
* Plasmodium falciparum malaria confirmed in blood smear
* Fever within the last 24 hours.

Exclusion Criteria:

* Treatment with an antimalarial agent within 72h of screening
* Severe concomitant disease
* Pregnant or breast-feeding women
* Women of child bearing potential not protected by an effective method of birth control

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Combination of fever clearance, general condition improvement at 48h parasite reduction at 72h and no need for rescue therapy at 72h | 3 initial days

SECONDARY OUTCOMES:
Parasite reduction | 3 initial days (72h)
Safety assessment | 28 days post 1st study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (4):
- Sanofi-Aventis Administrative Office, Porto-Novo, Benin
- Sanofi-Aventis Administrative Office, Ouagadougou, Burkina Faso
- Sanofi-Aventis Administrative Office, Libreville, Gabon
- Sanofi-Aventis Administrative Office, Dodoma, Tanzania

REFERENCES:
- [Derived] Held J, Supan C, Salazar CLO, Tinto H, Bonkian LN, Nahum A, Sie A, Abdulla S, Cantalloube C, Djeriou E, Bouyou-Akotet M, Ogutu B, Mordmuller B, Kreidenweiss A, Siribie M, Sirima SB, Kremsner PG. Safety and efficacy of the choline analogue SAR97276 for malaria treatment: results of two phase 2, open-label, multicenter trials in African patients. Malar J. 2017 May 4;16(1):188. doi: 10.1186/s12936-017-1832-x. PMID 28472957